CLINICAL TRIAL: NCT06553625
Title: Radiofrequency (RF) Ablation Prospective Outcomes Study for Central Nervous System
Brief Title: Radiofrequency (RF) Ablation Prospective Outcomes Study for Central Nervous System - RAPID for CNS
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: A4106; 92802182 (Other: Boston Scientific Corporation Protocol ID)
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease; Dystonia; Essential Tremor; Movement Disorders
MeSH Terms: conditions — Parkinson Disease; Dystonia; Essential Tremor; Movement Disorders | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Boston Scientific Radiofrequency Ablation Systems: Subjects treated with Boston Scientific commercially approved radiofrequency (RF) ablation systems in the central nervous system (CNS).
  Interventions: Device: Radiofrequency Ablation

INTERVENTIONS:
Device: Radiofrequency Ablation — Radiofrequency Ablation used in the central nervous system (CNS) in functional neurosurgery

SUMMARY:
The objective of this study is to compile real-world outcomes of Boston Scientific commercially approved radiofrequency (RF) ablation systems used in the central nervous system (CNS) for use in functional neurosurgery.

DETAILED DESCRIPTION:
The objective of this study is to compile real-world outcomes of Boston Scientific Corporation commercially approved radiofrequency (RF) ablation systems used in the central nervous system (CNS) for use in functional neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Study candidate is scheduled to be treated with a commercially approved Boston Scientific RF system for pain or for CNS applications per local Directions for Use (DFU)
* Signed a valid, IRB/EC/REB-approved informed consent form

Exclusion Criteria:

* Meets any contraindications per locally applicable Directions for Use (DFU)
* Currently diagnosed with cognitive impairment, or exhibits any characteristic, that would limit study candidate's ability to assess pain relief or to complete study assessments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients planned to receive treatment with a commercially approved Boston Scientific RF system to create lesions in the central nervous system (CNS) for use in functional neurosurgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Change in patient's quality of life (QoL) during the study as compared with baseline | Up to 24-Months
  Change in quality of life assessments during the study as compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Natalie M Bloom Lyons, M.A., Study Director — Boston Scientific Corporation
Locations (4):
- Germany (3):
  - Uniklinik Köln, Cologne
  - Universitaetsklinikum Dusseldorf, Düsseldorf
  - Universitaetsklinikum Wuerzburg, Würzburg
- St. Georges Hospital, London, United Kingdom